CLINICAL TRIAL: NCT02976337
Title: Effect of High-dose Target-controlled Naloxone Infusion on Pain and Hyperal-gesia in Patients Following Recovery From Impacted Mandibular Third Molar Extraction. A Randomized, Placebo-controlled, Double-blind Crossover Study.
Brief Title: Effect of High-dose Naloxone Following Third Molar Extraction
Acronym: TME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: mads u werner (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, mads u werner, Associate professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-15018869-TME
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Healthy Subjects; Hyperalgesia; Inflammations, Endodontic; Pain, Acute; Sensitization, Central
Keywords: Central sensitization; Endogenous opioids; Humans; Latent sensitization; Mandibular third molar extraction; Naloxone; Pain; Pressure algometry; Randomized controlled trial; Secondary hyperalgesia; Target controlled infusion
MeSH Terms: conditions — Hyperalgesia; Pulpitis; Acute Pain; Pain | interventions — Naloxone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose naloxone (Experimental): Naloxone 4 mg/ml i.v. infusion, total 3.25 mg/kg, target controlled infusion with three infusion rates (0.25 mg/kg; 0.75 mg/kg; 2.25 mg/kg) each of 25 min duration)
  Interventions: Drug: Naloxone
- Normal saline (Placebo Comparator): 0.9% physiological saline, i.v. infusion, total 0.81 ml/kg, target controlled infusion with three infusion rates (0.06 ml/kg; 0.19 ml/kg; 0.56 ml/kg) each of 25 min duration.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Naloxone — active drug infusion
  Other Names: Naloxon "B. Braun"
  Arms: High-dose naloxone
Drug: Normal Saline — placebo comparator
  Other Names: Physiologic Saline
  Arms: Normal saline

SUMMARY:
Recent studies have focused on the role of endogenous opioids on central sensitization. Central sensitization is known to be impaired or altered in chronic pain conditions, as fibromyalgia or chronic tension headache.

Animal studies have shown reinstatement of mechanical hypersensitivity following naloxone administration after resolution of an injury. This suggests latent sensitization. In the present study, the investigators hypothesize that a high-dose target-controlled naloxone infusion (total dose: 3.25 mg/kg) can reinstate pain and hyperalgesia 6-8 weeks after a unilateral primary open groin hernia repair procedure. The investigators aim to show that latent sensitization is present in humans and is modulated by endogenous opioids.

DETAILED DESCRIPTION:
Naloxone is a combined mu-opioid-receptor (MOR) inverse agonist and antagonist drug, which dose-dependently demonstrates hypoalgesic and hyperalgesic properties. Systemically administrated naloxone (3.0-10.0 mg/kg) and naltrexone (0.3-3.0 mg/kg) have been used in rodents to study the role of endogenous opioids on central processing of pain. It has been hypothesized that the endogenous opioid modulation of pain is impaired or altered in chronic pain conditions. Administration of naloxone and naltrexone following resolution of an inflammatory injury, have demonstrated a reinstatement of hypersensitivity to noxious stimuli, indicating a demasking of latent sensitization. It has thus been speculated that the endogenous opioid system may play an important role in the transition of acute to chronic pain in humans.

In an early human study using an electrical pain model, naloxone (21 microg/kg) increased the established area of secondary hyperalgesia (a measure of central sensitization).

In a previous translational placebo-controlled, double-blind, randomized, cross-over study in healthy humans, the investigators were unable to show naloxone-induced reinstatement of secondary hyperalgesia after resolution of a first-degree burn-injury (BI; H-2-2012-036). The investigators hypothesized, that the negative results were attributable to the low dose of naloxone (21 microg/kg) or perhaps insufficient tissue injury to generate latent sensitization.

The investigators therefore in a sequel study administered a higher dose of naloxone (2 mg/kg) 7 days after induction of a BI. The investigators demonstrated in 4 out of 12 subjects reinstatement of secondary hyperalgesia. The magnitude of reinstatement was more pronounced in high-sensitizers (subjects developing large secondary hyperalgesia areas immediately after the BI) The aims of the present clinical study in patients are first, to replicate our previous findings of naloxone-induced (3.25 mg/kg) unmasking of latent sensitization utilizing the impacted mandibular third molar extraction (TME) model with a more pronounced tissue injury than the BI-model. The endpoints are reinstatement of pain and hyperalgesia in the resolution-phase, 4 - 5 weeks after TME-surgery. Second, the study examines a potential dose-response relationship between three stable naloxone concentrations acquired by target controlled infusion (TCI).

ELIGIBILITY:
INCLUSION CRITERIA:

* Healthy male
* Age, minimum 18 yrs and maximum 65 yrs
* Signed informed consent
* Participants submitted to unilateral, primary, impacted, uncomplicated mandibular third molar extraction 4 weeks (+ 3 days) prior to examination Day 1.
* Standardized surgical procedure.
* Urin-sample without traces of opioids (morphine, methadon, buprenorphine, codeine, tramadol, ketobemidone, oxycodone, hydromorphone, dextromethorphan)
* ASA I-II
* Body mass index (BMI): 18 < BMI < 30 kg/m2

EXCLUSION CRITERIA:

* Participants, who do not speak or understand Danish
* Participants, who cannot cooperate with the investigation
* Participants, who have had previous surgery in the mandibular region
* Participants with pain at rest > 3 (NRS [0: no pain; 10: worst perceivable pain])
* Activity-related pain in the surgical field > 5 (NRS)
* Allergic reaction against morphine or other opioids (including naloxone),
* Abuse of alcohol or drugs - according to investigator's evaluation
* Use of psychotropic drugs (exception of SSRI)
* Neurologic or psychiatric disease
* Chronic pain condition
* Regular use of analgesic drugs
* Skin lesions or tattoos in the assessment areas
* Nerve lesions in the assessment sites (e.g., after trauma, dental surgery)
* Use of prescription drugs one week before the trial
* Use of over-the-counter (OTC) drugs 48 hours before the trial

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Change in the composite measure of pain (numerical rating scale (NRS); 0 = no pain; 10 = worst perceivable pain) | 1st session: 4 weeks after TME-surgery; 2nd session: 1 week later. At each session assessments are made at: -20 to -8 min; 15 to 25 min (TCI-step 1); 40 to 50 min (TCI-step 2); and 65 to 75 min (TCI-step 3) relative to start of TCI.
  during rest + masticatory pain + pain during external algometry (100 kPa) at the injury site

SECONDARY OUTCOMES:
Secondary hyperalgesia/allodynia area at mandibular skin sites directly overlying surgical and contralateral side | 1st session: 4 weeks after TME-surgery; 2nd session: 1 week later. At each session assessments are made at: -20 to -8 min; 15 to 25 min (TCI-step 1); 40 to 50 min (TCI-step 2); and 65 to 75 min (TCI-step 3) relative to start of TCI.
  Hyperalgesia/allodynia assessments with nylon monofilament (nominal value 4.93 [bending force: mean +/- SD = 69 +/- 14 mN]
Online Reaction Time | 1st session: 4 weeks after TME-surgery; 2nd session: 1 week later. At each session assessments are made at: -20 to -8 min; 15 to 25 min (TCI-step 1); 40 to 50 min (TCI-step 2); and 65 to 75 min (TCI-step 3) relative to start of TCI.
  measured using http://getyourwebsiteherecom/jswb/rttest01.htm. This computer-application shows a red-green traffic light. Participants are instructed to press the button when the light changes from red to green. Three measurements are used and the median value is used as a representative estimate of reaction time.
Hospital Anxiety and Depression Scale (HADS) | 1st session: 4 weeks after TME-surgery; 2nd session: 1 week later. Only pre-infusion
  HADS is used to assess anxiety and signs of depression. Based on 14 questions about the subject's status in the previous week, HADS measures agitation/anxiety and depression via two subscales (each containing seven questions). Participants have to answer each question on a scale of 0 to 3. The two subscales are summed separately. The maximum score of each subscale is 21 points and a score of 11 or more points suggests that the participant might be suffering from anxiety or depression. In case of score > 11 points in the depression subscale of the HADS, a physician will decide if there are clinical signs of depression. If there are signs of depression, this diagnosis will be told to the participant. The participant will be informed that the diagnosis of depression is based on clinical assessments - the HADS scale can be included in the diagnostic procedure. If it is the participants wish, he should visit his general practitioner for diagnosis and eventual treatment.
Pain Catastrophizing Scale (PCS) | 1st session: 4 weeks after TME-surgery; 2nd session: 1 week later. Only pre-infusion
  PCS consists of 13 questions divided into three sections: rumination, exaggeration and helplessness. The questions are answered in accordance to a scale of 0 to 4. There is evidence of catastrophizing thoughts at a total score > 30 points.
Clinical Opiate Withdrawal Scale (COWS) | 1st session: 4 weeks after TME-surgery; 2nd session: 1 week later. At each session assessments are made at: -20 to -8 min; 15 to 25 min (TCI-step 1); 40 to 50 min (TCI-step 2); and 65 to 75 min (TCI-step 3) relative to start of TCI.
  The Clinical Opiate Withdrawal Scale (COWS) is an examiner-based scale evaluating signs of opioid-withdrawal. Grading of symptoms, i.e. heart rate changes, sweating, restlessness, pupil size, bone or joint aches, running nose or tearing, nausea, vomiting, diarrhea, tremor, yawning, anxiety or irritability and "goose-flesh", are made in 11 categories. COWS-scores are divided into: 5-12 = mild; 13-24 = moderate; 25-36 = moderately severe ;> 36 = severe withdrawal reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Mads U Werner, MD, DMSc, Principal Investigator — Neuroscience Center, Copenhagen University Hospital, Denmark; Bradley K Taylor, M.Sc., Ph.D., Study Chair — Department of Physiology, University of Kentucky Medical Center
Locations (1):
- Neuroscience Center, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available as a supplementum to the published scientific article. Anticipated available in Spring 2018.

REFERENCES:
- [Background] Brennum J, Kaiser F, Dahl JB. Effect of naloxone on primary and secondary hyperalgesia induced by the human burn injury model. Acta Anaesthesiol Scand. 2001 Sep;45(8):954-60. doi: 10.1034/j.1399-6576.2001.450806.x. PMID 11576045
- [Background] Pielsticker A, Haag G, Zaudig M, Lautenbacher S. Impairment of pain inhibition in chronic tension-type headache. Pain. 2005 Nov;118(1-2):215-23. doi: 10.1016/j.pain.2005.08.019. Epub 2005 Oct 3. PMID 16202520
- [Background] Price DD, Staud R, Robinson ME, Mauderli AP, Cannon R, Vierck CJ. Enhanced temporal summation of second pain and its central modulation in fibromyalgia patients. Pain. 2002 Sep;99(1-2):49-59. doi: 10.1016/s0304-3959(02)00053-2. PMID 12237183
- [Background] van Wilgen CP, Keizer D. The sensitization model to explain how chronic pain exists without tissue damage. Pain Manag Nurs. 2012 Mar;13(1):60-5. doi: 10.1016/j.pmn.2010.03.001. Epub 2010 Jul 22. PMID 22341140
- [Result] Koppert W, Filitz J, Troster A, Ihmsen H, Angst M, Flor H, Schuttler J, Schmelz M. Activation of naloxone-sensitive and -insensitive inhibitory systems in a human pain model. J Pain. 2005 Nov;6(11):757-64. doi: 10.1016/j.jpain.2005.07.002. PMID 16275600
- [Result] Campillo A, Cabanero D, Romero A, Garcia-Nogales P, Puig MM. Delayed postoperative latent pain sensitization revealed by the systemic administration of opioid antagonists in mice. Eur J Pharmacol. 2011 Apr 25;657(1-3):89-96. doi: 10.1016/j.ejphar.2011.01.059. Epub 2011 Feb 4. PMID 21300053
- [Result] Taylor BK, Corder G. Endogenous analgesia, dependence, and latent pain sensitization. Curr Top Behav Neurosci. 2014;20:283-325. doi: 10.1007/7854_2014_351. PMID 25227929
- [Result] Corder G, Doolen S, Donahue RR, Winter MK, Jutras BL, He Y, Hu X, Wieskopf JS, Mogil JS, Storm DR, Wang ZJ, McCarson KE, Taylor BK. Constitutive mu-opioid receptor activity leads to long-term endogenous analgesia and dependence. Science. 2013 Sep 20;341(6152):1394-9. doi: 10.1126/science.1239403. PMID 24052307
- [Result] Pereira MP, Werner MU, Ringsted TK, Rowbotham MC, Taylor BK, Dahl JB. Does naloxone reinstate secondary hyperalgesia in humans after resolution of a burn injury? A placebo-controlled, double-blind, randomized, cross-over study. PLoS One. 2013 May 31;8(5):e64608. doi: 10.1371/journal.pone.0064608. Print 2013. PMID 23741350
- [Result] Pereira MP, Donahue RR, Dahl JB, Werner M, Taylor BK, Werner MU. Endogenous Opioid-Masked Latent Pain Sensitization: Studies from Mouse to Human. PLoS One. 2015 Aug 25;10(8):e0134441. doi: 10.1371/journal.pone.0134441. eCollection 2015. PMID 26305798
- [Result] Edwards RR, Ness TJ, Fillingim RB. Endogenous opioids, blood pressure, and diffuse noxious inhibitory controls: a preliminary study. Percept Mot Skills. 2004 Oct;99(2):679-87. doi: 10.2466/pms.99.2.679-687. PMID 15560360
- [Result] Singla NK, Desjardins PJ, Chang PD. A comparison of the clinical and experimental characteristics of four acute surgical pain models: dental extraction, bunionectomy, joint replacement, and soft tissue surgery. Pain. 2014 Mar;155(3):441-456. doi: 10.1016/j.pain.2013.09.002. Epub 2013 Sep 6. PMID 24012952
- [Result] Glass PS, Jhaveri RM, Smith LR. Comparison of potency and duration of action of nalmefene and naloxone. Anesth Analg. 1994 Mar;78(3):536-41. doi: 10.1213/00000539-199403000-00021. PMID 8109774